CLINICAL TRIAL: NCT04762914
Title: Observing the Perioperative Effects of Prehabilitation in Colorectal Cancer
Brief Title: Observing the Perioperative Effects of Prehabilitation in Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Medway Primary Care Trust (Other Government)
Responsible Party: Principal Investigator, Richard Dickson-Lowe, Consultant Surgeon, Medway Primary Care Trust
Other Study IDs: 2021.038N
Record Dates: First submitted 2021-01-22; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Colon Cancer
Keywords: Prehabilitation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation (PH): Patients who underwent prehabilitation prior to colorectal cancer resection
  Interventions: Other: Prehabilitation
- Non-Prehabilitation (NPH): Patients who did not undergo prehabilitation prior to colorectal cancer resection

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation is a multimodal and multidisciplinary person-centred perioperative approach involving supervised exercise training, nutritional education, management of polypharmacy and psychological advice.
  Groups: Prehabilitation (PH)

SUMMARY:
Quality Improvement Project to evaluate how prehabilitation can be incorporated into our colorectal cancer pathway and assess its clinical benefits.

DETAILED DESCRIPTION:
The aim was to evaluate how prehabilitation (PH) can be incorporated into our colorectal cancer pathway and assess its clinical benefits.

Patients underwent PH (exercise, nutrition and psychological support) before resection of colorectal carcinoma in a DGH over fourteen months. Patients were matched by operation, age, sex and ASA to non-prehabilitation (NPH) patients using a prospectively maintained database. Length of stay (LoS) and complication rate and 90-day readmission rates were compared using Wilcoxon and McNemar's methods.

Prehabilitation significantly improved peak VO2 and AT. This corresponds to a reduction in predicted 30-day mortality. Despite a higher Charlson index LoS was unchanged suggesting prehabilitation may permit safe resection in comorbid patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 who had prehabilitation for colorectal cancer

Exclusion Criteria:

* Children
* Patients who had prehabilitation but not for colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients over the age of 18 needing surgery were identified from clinics, endoscopy or weekly multidisciplinary meetings (MDT). Patients who were clinically judged to be frail or had multiple comorbidities were referred for prehabilitation prior to resection. Those that underwent prehabilitation were matched using operation type, age, sex and ASA with patients who did not have prehabilitation prior to resection. Surgery for all patients was carried out within the context of an enhanced recovery programme.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | From date of operation to date of discharge in number of days over a 90 day follow up period
  Time spent in hospital
Complication rate | Follow up over a period of 90 days following operation
  All Clavien-Dindo complications

SECONDARY OUTCOMES:
Anaerobic threshold | CPET performed before prehabilitation and after prehabilitation (median of 36 days)
  Measured by looking at CPET results pre- and post- prehab

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Dickson-Lowe, Principal Investigator — Medway PCT
Locations (1):
- Medway Hospitals NHS Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No